CLINICAL TRIAL: NCT04577300
Title: A Randomized, Sham Controlled, Masked Phase II Study to Evaluate the Safety and Efficacy of Dual Intravitreal Implantation of NT-501 Encapsulated Cell Therapy for the Treatment of Glaucoma
Brief Title: Dual Intravitreal Implantation of NT-501 Encapsulated Cell Therapy for Glaucoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 56950
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dual Implantation (Experimental): Two NT-501 devices will be implanted in the study eye.
  Interventions: Drug: NT-501
- Single Implantation (Experimental): One NT-501 device will be implanted in the study eye.
  Interventions: Drug: NT-501
- Sham Implantation (Sham Comparator): No NT-501 devices will be implanted in the study eye.
  Interventions: Other: Sham comparator

INTERVENTIONS:
Drug: NT-501 — Implant of Neurotech NT-501 device(s)
  Arms: Dual Implantation; Single Implantation
Other: Sham comparator — Sham implantation
  Arms: Sham Implantation

SUMMARY:
To determine the safety and efficacy over 24 months of dual NT-501 CNTF encapsulated cell therapy (ECT) on visual impairment related to glaucoma.

DETAILED DESCRIPTION:
A randomized, sham controlled, masked trial of up to 30 eyes will be recruited into the study. Participants with a qualifying study eye will be randomized after screening and baseline evaluations to receive 2 NT-501 ECT implants in the study eye (20 eyes), 1 NT-501 ECT implant (5 eyes) or a sham surgery (control arm; 5 eyes). No explant will be required. An examination for safety will occur one day and one week following implant and periodically thereafter for 24 months post-implant. Patients in the control arm may be offered 2 NT-501 ECT implants after the 12-month post-operative follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be medically able to undergo the testing required in the schedule of events (SOE).
2. Participant's clinical diagnosis must be consistent with glaucoma characterized by the following features: Mean deviation (MD) of -3 to -20 dB on Humphrey Visual Field 24-2 testing and two visual field tests of adequate quality with a maximum VFI variability of ± 10%
3. Residual visual field preservation including best-corrected visual acuity (BCVA) better than 20/200 in either eye.
4. Participant's eye pressure must be clinically stable, with IOP <21.
5. If a participant has two eyes meeting study criteria, the worse eye as determined by visual field index (VFI) or patient preference, will be deemed includable. If both eyes qualify and have the same VFI, a randomization procedure will assign one eye to the study.
6. Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.
7. Females of childbearing potential must agree to use an effective form of birth control.
8. Participant must be determined by the presurgical anesthesia or medical team to be fit for ophthalmic surgery for the NT-501 ECT implant insertion.

Exclusion Criteria:

1. Participant is unable to comply with study procedures or followup visits.
2. Participant has other optic nerve or retinal degenerative disease causing vision loss, irrespective of whether it is currently treated or untreated.
3. Participant is likely to be offered glaucoma surgery in the study eye within 6 months of screening.
4. Participant has cataract-associated vision loss to less than 20/40.
5. Participant has a history of ocular herpes zoster.
6. Participant has a requirement of acyclovir and/or related products during study duration. To be eligible for this study, the participant must discontinue use of these products prior to enrollment and must not continue with the products until after they have completed the study.
7. Participant has evidence of corneal opacification or lack of optical clarity.
8. Participant has uveitis or other ocular inflammatory disease.
9. Participant is receiving systemic steroids or other immunosuppressive medications.
10. Participant has diabetic macular edema and/or diabetic retinopathy.
11. Participant has myopic degeneration.
12. Participant is currently participating in or has within the last 3 months participated in any other clinical trial of a drug by ocular (if in the study eye) or systemic administration.
13. Participant is pregnant or lactating.
14. Participant is on chemotherapy.
15. Participant has a history of malignancy other than basal cell carcinoma, unless it was treated successfully 2 years prior to inclusion in the trial.
16. Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments.
17. Any intraocular surgery of the study eye within 12 weeks prior to the screening visit
18. History of use of drugs with known retinal toxicity, at retinotoxic doses.
19. Patient has a history of multiple sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Visual Field MD at 12 Months | 12 months
  Change from baseline in visual field through 12 months as assessed by Mean Deviation (MD).

SECONDARY OUTCOMES:
Visual Field Index at 12 months | 12 months
  Change from baseline in visual field through 12 months as assessed by Visual Field Index (VFI).
Visual Field PLR at 12 months | 12 months
  Change from baseline in visual field pointwise linear regression (PLR) through 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States